CLINICAL TRIAL: NCT00807781
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Mammaglobin-A DNA Vaccine in Breast Cancer Patients With Metastatic Disease
Brief Title: Mammaglobin-A DNA Vaccine for Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0298 / 201110267
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mammaglobin-A DNA vaccine (Experimental): Patients will receive vaccine day 1 (week 1), week 4 (day 29 +/- 7), week 8 (day 57 +/- 7) with at least 21 days between injection days.
  All injections will be given intramuscularly using a jet delivery device.
  Patients will be administered the vaccine in lateral shoulder and buttocks positions that will be rotated with each administration in the above order.
  Interventions: Biological: Mammaglobin-A DNA vaccine

INTERVENTIONS:
Biological: Mammaglobin-A DNA vaccine

SUMMARY:
The purpose of this study is to evaluate the safety of mammaglobin-A DNA vaccine in metastatic breast cancer patients.

DETAILED DESCRIPTION:
This is a phase I open-label study to evaluate the safety and immunogenicity of a plasmid mammaglobin-A DNA vaccine. The plasmid mammaglobin-A DNA vaccine will be formulated as a naked plasmid DNA vaccine (WUSM-MGBA-01). The hypothesis of this study is that the mammaglobin-A DNA vaccine will be safe for human administration and capable of generating measurable CD8 T cell responses to mammaglobin-A. The primary objective of this study is to demonstrate the safety of the mammaglobin-A DNA vaccine. The secondary objective is to evaluate the immunogenicity of the mammaglobin-A DNA vaccine as measured by ELISPOT analysis, a surrogate for CD8 T cell function.

ELIGIBILITY:
Inclusion Criteria

A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

* Patient must have a histologically confirmed diagnosis of invasive breast cancer. Paraffin-embedded tissue or tissue sections must be available for immunohistochemistry analysis to confirm mammaglobin-A expression.
* Patient must have metastatic breast cancer that has been stable for at least 30 days. This may include patients with measurable or evaluable disease by RECIST criteria, and those without evidence of disease.
* Patient must not have had chemotherapy, radiation therapy, or biologic therapy within 30 days of initiating therapy on study, and have resolved all toxicities experienced from these treatments. Patients receiving hormonal therapy and supportive therapy with bisphosphonates will be allowed. Patients currently on trastuzumab will be allowed.
* Patient must be 18 years or older.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient must have a life expectancy of ≥ 24 weeks.
* Patient must have adequate organ and marrow function as defined below:

  * WBC ≥3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * total bilirubin ≤2.5 X institutional upper limit of normal
  * AST/ALT ≤2.5 X institutional upper limit of normal
  * creatinine ≤1.5 X institutional upper limit of normal
* Women of reproductive potential must have a negative urine or serum β-HCG pregnancy test prior to enrollment to confirm that they are not pregnant.
* Women of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 21 days prior to study entry and for the duration of study participation (until Week 52).
* Patient must be available for follow-up through week 52 of the study.
* The patient with a previous history of non-breast malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patients have been considered disease free for at least 1 year (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix)
* Patient must be able and willing to sign a written informed consent document.

Exclusion Criteria

A patient will be ineligible for inclusion in this study if ANY of the following criteria apply:

* Patient has evidence of progressive breast cancer within the last 30 days.
* Patient is currently receiving other investigational agent(s) or has received an investigational agent within the last 30 days.
* Patient has known brain metastases.
* Patient with known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patient with prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Patient is pregnant.
* Patients known to be HIV-positive are ineligible because of the potential inability to generate an immune response to vaccines.
* Patients has failed greater than two chemotherapy regimens for metastatic disease.
* Subjects with a strong likelihood of non-adherence such as difficulties in adhering to follow-up schedule due to geographic distance from the Siteman Cancer Center, should not knowingly be registered.
* Patients who have known seropositivity for hepatitis B antigen or hepatitis C antibody. Testing will be done prior to study entry to confirm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of mammaglobin-A DNA vaccine, WUSM-MGBA-01 | 30 days after completion of treatment

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the mammaglobin-A DNA vaccine, WUSTL-MGBA-01. Immunogenicity will be measured by ELISPOT analysis, a surrogate for CD8 T cell function. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, M.D., Principal Investigator — Washington Univerisity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu